CLINICAL TRIAL: NCT07376720
Title: A Clinical Study Evaluating the Safety and Efficacy of BCMA-GPRC5D CAR-T in Patients With Relapsed/Refractory Multiple Myeloma Who Have Received Three or More Lines of Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Donghua Zhang (Other)
Responsible Party: Sponsor-Investigator, Donghua Zhang, professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHZ1962-G
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recurrent/refractory multiple myeloma (r/r MM) patients received infusion of BCMA-GPRC5D CAR-T cells (Experimental)
  Interventions: Drug: Recurrent/refractory multiple myeloma (r/r MM) patients received infusion of BCMA-GPRC5D CAR-T cells

INTERVENTIONS:
Drug: Recurrent/refractory multiple myeloma (r/r MM) patients received infusion of BCMA-GPRC5D CAR-T cells — Recurrent/refractory multiple myeloma (r/r MM) patients received infusion of BCMA-GPRC5D CAR-T cells

SUMMARY:
This research project includes patients with relapsed/refractory multiple myeloma (r/r MM) who have received more than three lines of treatment, including those with secondary recurrence, SCT recurrence, and refractory cases. Through this study, we aim to preliminarily determine the effectiveness of the treatment for r/r MM, with the expectation of providing new treatment methods to improve the survival rate of patients with r/r MM.

ELIGIBILITY:
Inclusion Criteria:

1. The patient or their guardian understands and voluntarily signs the informed consent form, and is expected to complete the follow-up examinations and treatments of the research procedures;
2. Age 18-75 years (inclusive), gender not limited;
3. According to the IMWG diagnostic criteria, patients diagnosed with multiple myeloma;
4. Based on any of the following criteria, measurable lesions are determined during the screening: the level of single-clonal paraprotein (M-protein) in the blood ≥ 1.0 g/dL or the M-protein level in urine ≥ 200 mg/24 hours; or a light chain-type multiple myeloma diagnosed as having no measurable lesions in serum or urine: the free light chain of serum immunoglobulin ≥ 10 mg/dL and the abnormal ratio of free light chains of serum immunoglobulin κ/γ;
5. Has received at least three lines of treatment for multiple myeloma in the past, and should include:

   1. One proteasome inhibitor (such as bortezomib, carfilzomib, ixazomib, etc.);
   2. One immunomodulator (such as thalidomide, lenalidomide, pomalidomide, etc.);
   3. One CD38 monoclonal antibody;
6. There is evidence that the patient's multiple myeloma disease is relapsed/refractory or primary refractory, defined as:

   1. Relapsed/refractory: no response to salvage therapy (no response is defined as not achieving minimal response [MR] or disease progression during treatment), or disease progression within 60 days after the last treatment, or disease progression after achieving MR or the above remission;
   2. Primary refractory: no MR or above treatment response has been achieved, including patients who have never achieved MR or above remission, but the M-protein has not changed significantly and there is no clinical progression evidence, and patients with primary refractory and progression, meeting the progression definition.
7. The patient has recovered from the toxicity of previous treatment, that is, the CTCAE toxicity grade is less than 2 (unless the abnormality is related to the tumor or is judged by the investigator to be in a stable state, which has little impact on safety or efficacy);
8. The ECOG performance status score is 0-2 and the estimated survival period is more than 3 months;
9. Has appropriate organ function:

   1. Alanine aminotransferase (ALT) ≤ 3 times the upper limit of normal value (ULN);
   2. Aspartate aminotransferase (AST) ≤ 3 times ULN;
   3. Total bilirubin ≤ 1.5 times ULN;
   4. Serum creatinine ≤ 1.5 times ULN, or creatinine clearance rate ≥ 60 mL/min;
   5. Hemoglobin ≥ 50g/L (must not have received blood transfusion support within 7 days before laboratory examination);
   6. Intraocular oxygen saturation ≥ 92%;
   7. Corrected serum calcium ≤ 12.5 mg/dL (≤ 3.1 mmol/L) or free ionized calcium ≤ 6.5 mg/dL (≤ 1.6 mmol/L);
   8. Left ventricular ejection fraction (LVEF) ≥ 45%, confirmed by echocardiography that there is no pericardial effusion, and no clinically significant electrocardiogram findings;
   9. No clinically significant pleural effusion;
10. The required venous access can be established, and there are no contraindications for white blood cell collection.

Exclusion Criteria:

1. Within 3 years, diagnosed with or treated for any other aggressive malignant tumor other than multiple myeloma;
2. Previously received the following anti-tumor treatments (before collecting and preparing the CAR-T cells): within 14 days or at least 5 half-lives (whichever is shorter) received targeted therapy, epigenetic therapy or experimental drug treatment, or used invasive experimental medical devices; received monoclonal antibody treatment for multiple myeloma within 21 days; received cytotoxic treatment within 14 days; received proteasome inhibitor treatment within 14 days; received immunomodulatory agent treatment within 7 days; received radiotherapy within 14 days (except for fields covering ≤5% of bone marrow reserves);
3. Suspected that MM has involved the central nervous system or meninges and confirmed by MRI or CT, or has other active central nervous system diseases;
4. At the screening stage, had Waldenström macroglobulinemia, POEMS syndrome (multiple neuropathy, organ enlargement, endocrine lesion, monoclonal protein disease and skin changes) or primary AL amyloidosis;
5. Positive for hepatitis B surface antigen (HBsAg), or positive for hepatitis B core antibody (HBcAb) and peripheral blood HBV DNA titer is higher than the lower limit set by the research institution; positive for hepatitis C virus (HCV) antibody and positive for peripheral blood HCV-RNA; positive for human immunodeficiency virus (HIV) antibody; quantitative detection of cytomegalovirus (CMV) DNA is higher than the lower limit set by the research institution; positive for syphilis spirochete antibody; quantitative detection of Epstein-Barr virus (EBV) DNA is higher than the lower limit set by the research institution;
6. Those with a history of severe allergic reactions [severe allergic reactions are defined as secondary or higher-level allergic reactions, and when allergic reactions occur, any of the following clinical manifestations occur: airway obstruction (runny nose, cough, wheezing, breathing difficulty), tachycardia, hypotension, arrhythmia, gastrointestinal symptoms (nausea, vomiting), incontinence of urine and stool, laryngeal edema, bronchospasm, cyanosis, shock, cardiac and respiratory arrest) or known to be sensitive to any active ingredients of the drugs included in this test, excipients, or murine products, or cross-reactive proteins from different species;
7. Suffering from severe heart diseases, including but not limited to severe arrhythmia, unstable angina pectoris,大面积 myocardial infarction， NYHA class III or IV cardiac insufficiency before screening， having had a myocardial infarction within ≤ 6 months before screening or having received coronary artery bypass grafting (CABG)， having a history of unexplained syncope not caused by vasovagal or dehydration， severe non-ischemic cardiomyopathy history， refractory hypertension (refractory hypertension is defined as： after improving lifestyle， using reasonable and tolerable sufficient ≥ 3 types of antihypertensive drugs (including diuretics) for more than 1 month， blood pressure still cannot be controlled or taking ≥ 4 types of antihypertensive drugs can effectively control blood pressure)；
8. Systemic diseases judged by the investigator to be unstable： including but not limited to severe liver， kidney or metabolic diseases requiring drug treatment；
9. Had acute/chronic graft-versus-host disease (GVHD) within 6 months before screening， or patients requiring immunosuppressive therapy for GVHD；
10. Patients with active autoimmune or inflammatory diseases of the nervous system (such as Guillain-Barré syndrome (GBS)， amyotrophic lateral sclerosis (ALS)) and clinically significant active cerebrovascular diseases (such as brain edema， posterior reversible encephalopathy syndrome (PRES))；
11. Those with tumor emergencies (such as spinal cord compression， intestinal obstruction， leukocyte stasis， tumor dissolution syndrome， etc.) requiring emergency treatment before screening or during reinfusion；
12. Have infections that require antibiotic treatment， such as uncontrolled bacterial， fungal， viral or other infections；
13. Within 1 week before blood collection for CAR-T preparation， have used drugs that affect the patient's blood count.

    Short-acting hematopoietic cytokine drugs, or those who have used long-acting hematopoietic cytokine drugs within 2 weeks and whose preparation has been affected by the study investigators.
14. During the screening, within 2 weeks before the planned preparation of CAR-T cells, those who are currently receiving hormones or immunosuppressive drugs, and whose preparation is judged to be affected by the study investigators:

    1. Hormones: Those who are currently receiving systemic steroid therapy and whose treatment requires long-term systemic steroid therapy during the treatment period (except for inhalation or local use); and those who received systemic steroid therapy within 72 hours before the cell infusion (except for inhalation or local use);
    2. Immunosuppressants: Those who are currently receiving immunosuppressants;
15. Within 4 weeks before the conditioning regimen, those who have undergone major surgery (except diagnostic surgery and biopsy) or those whose major surgery is planned during the study period, or those whose surgical wounds have not fully healed before enrollment;
16. Within 4 weeks before the screening, those who have received (attenuated) live virus vaccines;
17. Those with severe mental disorders;
18. Those who are heavy drinkers or have a history of drug abuse;
19. Pregnant or lactating women, and female subjects who plan to conceive within 2 years after the cell infusion or whose male partners plan to conceive within 2 years after the cell infusion;

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2028-10-30 (Estimated); Study Completion 2029-10-30 (Estimated)

PRIMARY OUTCOMES:
overall survival | 1,3,6,12,18,24 months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China